CLINICAL TRIAL: NCT03201601
Title: Comparison of the Effect of a Combination of Myoinositol:D-chiro-inositol With Low Proportion of DCI (40:1) Versus a Combination With a Higher Proportion of DCI (3.6:1) in the Oocyte Quality and Pregnancy Rates in Women With PCOS
Brief Title: Evaluation of the Mixture Myoinositol:D-chiro-inositol 3.6:1 in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C015
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2016-10

CONDITIONS: Polycystic Ovarian Syndrome; Infertility
Keywords: Polycystic ovarian syndrome; D-chiro-inositol; Fertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Inositol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 550 mg of MYO and 150 mg of DCI (Experimental): Volunteers will take twice at day for 12 weeks a capsule containing 550 mg of myo-inositol and 150 mg of D-chiro-inositol.
  Interventions: Drug: D-chiro-inositol; Drug: Myoinositol
- 550 mg of MYO and 13.8 mg of DCI (Active Comparator): Volunteers will take twice at day for 12 weeks a capsule containing 550 mg of myo-inositol and 13.8 mg of D-chiro-inositol.
  Interventions: Drug: D-chiro-inositol; Drug: Myoinositol

INTERVENTIONS:
Drug: D-chiro-inositol — Each participant will consume 2 capsules daily of each treatment, in the morning and at night without any restriction in the diet nor in their habits of life. The treatment will last 12 weeks.
  Other Names: Cis-1,2,4-trans-3,5,6-cyclohexanehexol
Drug: Myoinositol — Each participant will consume 2 capsules daily of each treatment, in the morning and at night without any restriction in the diet nor in their habits of life. The treatment will last 12 weeks.
  Other Names: cis-1,2,3,5-trans-4,6-cyclohexanehexol

SUMMARY:
The aim of the present study is to evaluate the effect of increasing the proportion of D-chiro-inositol (DCI) in a combination with myo-inositol (MYO) in improving fertility in women with polycystic ovarian syndrome (PCOS). Sixty women diagnosed with PCOS will randomly take twice a day for 12 weeks a capsule containing 550 mg of myo-inositol and 150 mg of D-chiro-inositol or capsules containing 550 mg of myo-inositol and 13.8 mg of D-chiro-inositol.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is the most prevalent endocrinopathy in women of childbearing age. It affects 4-8% of the population and of them, approximately 74% present anovulatory cycles and, therefore, fertility problems.

Both myo-inositol and D-chiro-inositol are 2 natural substances that have been shown to improve ovarian function and metabolism in women with polycystic ovarian syndrome.

The aim of the present study is to compare the effect of 2 ratios of myo-inositol /D-chiro-inositol on parameters related to the fertility of women with PCOS.

It is a multicenter, controlled, randomized, double-blind, parallel-group, 12-week clinical trial which will be conducted in 13 public and private hospitals from Spain.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with PCOS according to Rotterdam criteria.
* Being in in vitro fertilization treatment.
* Body mass index less than 30 kg/m2.
* Accept freely to participate in the study and sign the informed consent document.

Exclusion Criteria:

* Contraindication to perform techniques of assisted reproduction or stimulation of ovulation.
* Advanced state of endometriosis (III or IV).
* Classified as poor responder in fertility treatment.
* Premature ovarian failure.
* Severe male factor (cryptozoospermia).
* Few expectations of compliance and/or collaboration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 12 weeks
  Number of pregnancies

SECONDARY OUTCOMES:
Mature MII oocytes | 12 weeks
  Number of mature MII oocytes
IM/VG oocytes | 12 weeks
  Number of IM/VG oocytes
Grade I, II, III embryos | 12 weeks
  Number of embryos of degree I, II, III
Days of stimulation | 12 weeks
  Days of stimulation
Gestational sacs | 12 weeks
  Number of gestational sacs
Transferred embryos | 12 weeks
  Number of embryos transferred
Total testosterone | 12 weeks
  Total testosterone levels
Glucose | 12 weeks
  Glucose levels
Insulin | 12 weeks
  Insulin levels

CONTACTS AND LOCATIONS:
Overall Officials: Nicolás Mendoza, MD, PhD, Principal Investigator — Professor of Gynecology at the Faculty of Medicine of the University of Granada

IPD SHARING:
Plan to Share IPD: No